CLINICAL TRIAL: NCT03918954
Title: Comparison of Physical and Virtual Sensory Room in an Inpatient Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Stockholm University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: VGRVR
Record Dates: First submitted 2019-01-10; First posted 2019-04-18 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2020-06

CONDITIONS: Anxiety State; Depression; Bipolar Depression
MeSH Terms: conditions — Anxiety Disorders; Depression; Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical sensory room (Active Comparator): In the inpatient ward there is a specifically designed room for calming down which a patient can request access to. In the room there is calming music, soft mats, nature themed wallpaper and calming visual lighting.
  Interventions: Other: Sensory room
- Virtual sensory room (Experimental): The patients will have access to wireless virtual reality glasses during a session. The glasses will have a specially made protection that will be disinfected between each user, all users will also have the opportunity to choose a disposable cover for the glasses. The VR glasses are adjustable and adaptable to all types of head sizes and can be used with regular glasses. The application accessable in the VR glasses is called Calm Place, a virtual natural environment with day and night cycles, dynamic weather and associated soundscapes.
  Interventions: Device: Virtual sensory room

INTERVENTIONS:
Device: Virtual sensory room — A pair of virtual reality glasses (Oculus Go) with installed the program Calm Place, a program designed for anxiety reduction.
  Arms: Virtual sensory room
Other: Sensory room — A room with calming elements that patients can use to feel calm.
  Arms: Physical sensory room

SUMMARY:
Sensory room is a new method in psychiatric inpatient care for management of anxiety. Since this method for anxiety management is being implemented more and more extensively within the psychiatric care system it is important to study its effect and whether there is any difference between physical and virtual sensory.

In this study, the effect on mental well-being, pulse and blood pressure will be compared before and after each use of a virtual or physically sensory room. How the different methods affect the total care time, use of anxiety medication and results from self-assessment scales to measure depression and anxiety symptoms will also be looked at. The study will be conducted on two separate wards which primarily care for patients with the primary diagnosis of bipolar disorder.

DETAILED DESCRIPTION:
This study will include about 100 research subjects admitted to an inpatient ward at the department of psychiatry for affective disorder. The study will be conducted in two inpatient wards. Patients who consent to participation will be offered to stay in a sensory room (a physical sensory room in one ward and a virtual sensory room via a pair of wireless VR glasses in another ward). In connection with the use of the virtual or physical sensory room, the patients will be given a visual analogue scale which asks the patient to rate their overall anxiety and mental health on a scale from 1 (feeling very bad) to 10 (feeling excellent). This will be the primary measure of the study. Before and after each visit the participant will have their pulse and blood pressure measured.

Included patients will also be asked about participation in individual interviews. Semi-structured interviews will be carried out and collected data will be analyzed with a phenomenological approach. The purpose of this study is to shed light on experiences of staying in the digital and analogue sensory rooms.

A number of self-rated questionnaires will be used in the project to establish the research subjects' level of depression and anxiety during their inpatient stay.

* The Montgomery-Åsberg Depression Rating (MADRS-S) scale. MADRS-S is a self-assessment tool for assessing depression symptoms, it is used regularly in the clinic to evaluate depression symptoms. The inventory consists of a self-assessment form containing 9 statements intended to measure different depression symptoms. This scale is administered at the enrollment interview if patient consents to participation and once weekly until discharge.
* Beck Anxiety Inventory (BAI) is a self-assessment instrument that measures the degree of anxiety. The inventory consists of a self-assessment form containing 21 statements intended to measure 21 different anxiety symptoms. This scale is administered at the enrollment interview if patient consents to participation and once weekly until discharge.
* The Clinical Global Impressions (CGI) scale. CGI is a 7-scaled evaluation tool that requires the physician to determine the degree of the patient's disease at the time of assessment, in relation to the clinician's previous experience in patients with the same diagnosis. This scale is administered at the enrollment interview if patient consents to participation and once weekly until discharge.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to one of the two eligible inpatient units
* Age over 18 years

Exclusion Criteria:

* Diagnosis of schizophrenia (ICD-10 F20) or schizoaffective disorder (ICD-10 F25)
* Intellectual developmental disorder, organic brain injury or other condition that precludes informed consent
* Active withdrawal symptoms from alcohol or other substances of abuse
* Visual or balance disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Change on Visual Analogue Scale of anxiety | Immediately before and following the first administration of treatment
  A visual analogue scale from 0 (lowest) to 10 (highest) level of anxiety

SECONDARY OUTCOMES:
Beck´s Anxiety Scale | Once weekly from date of inclusion until the date of discharge up to 3 weeks
  Total score on 21 self-rated questions on anxiety (ranging from 0=no anxiety to 63=maximum level of anxiety)
Montgomery-Åsberg Depression Rating Scale (MADRS-S) | Once weekly from date of inclusion until the date of discharge up to 3 weeks
  Depression grade on a self-rating scale ranging from 0=no depression to 54=most severe depression
Use of anxiolytic medication | Total use of medication from date of inclusion to date of discharge up to 3 weeks
  Use in mg of anxiolytic medication
Clinical Global Impression | Once weekly from date of inclusion until the date of discharge up to 3 weeks
  Clinician assessment of patient´s overall mental state ranging from 0 (no symptoms) to 7 (severe mental illness)
Length of stay | Length of admission in days from date of inclusion to date of discharge up to a year
  Number of days admitted to inpatient care
Blood pressure | Immediately before and following first administration of treatment
  mmHg before and after intervention
Pulse | Immediately before and following first administration of treatment
  Heartbeats per minute before and after intervention
Visual Analogue Scale of anxiety | An average of each immediate before and following measure of the administration of treatment
  A visual analogue scale from 0 (lowest) to 10 (highest) level of anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Steinn Steingrimsson, PhD, Study Director — Sahlgrenska Academy
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ilioudi M, Lindner P, Ali L, Wallstrom S, Thunstrom AO, Ioannou M, Anving N, Johansson V, Hamilton W, Falk O, Steingrimsson S. Physical Versus Virtual Reality-Based Calm Rooms for Psychiatric Inpatients: Quasi-Randomized Trial. J Med Internet Res. 2023 May 19;25:e42365. doi: 10.2196/42365. PMID 37204858